CLINICAL TRIAL: NCT03955237
Title: Perioperative Fluid Management According to the Preoperative and Perioperative Glucose
Brief Title: Perioperative Fluid Management According to the Preoperative and Perioperative Glucose Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayse Cigdem Tutuncu, Assoc Prof, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 82546
Record Dates: First submitted 2017-08-20; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Perioperative Complication

STUDY DESIGN:
Intervention Model Description: 3 different type of fluid

ARMS (3):
- non glucose infusion group (Active Comparator): Drug: LR infusion LR solution without glucose; the patients with preoperative blood glucose level higher than 90 mg/dL.
  Interventions: Procedure: Drug: dextrose containing infusion
- Drug:1% Dextrose infusion group (Active Comparator): Drug:LR+ 1% Dextrose infusion LR solution with % 1 glucose: the patients with preoperative blood glucose level between 60-90 mg/dL,
  Interventions: Procedure: Drug: dextrose containing infusion
- 2% Dextrose infusion group (Active Comparator): Drug:LR+ 2 % Dextrose infusion Lactate ringer (LR) solution with % 2 glucose; the patients with preoperative blood glucose level lower than 60 mg/dL,
  Interventions: Procedure: Drug: dextrose containing infusion

INTERVENTIONS:
Procedure: Drug: dextrose containing infusion — Drug: infusing dextrose containing or non glucose fluid according to blood glucose level
  Other Names: drug: non dextrose containing infusion

SUMMARY:
Background:Hyperglycemia and hypoglycemia both cause detrimental side effects for pediatric patients. Prolonged fasting time, age dependent physiological diffences and individual differences of patients make complicated the perioperative fluid therapy. Isotonic electrolyte solutions without glucose or with lower glucose concentrations recommended for intraoperative period in pediatric patients.

Objective: The aim of this prospective study is to evaluate the different glucose concentrations(without dextrose, 1 % dextrose+LR, 2 % dextrose+LR) in perioperative infusion solutions according to preoperative blood glucose level to maintain normoglycemia in pediatric patients.

Method: The consecutive 250 eligible pediatric patients aged between 6 months- 12 years with ASA risk score of I-II undergoing surgery lasting less than four hours were enrolled the study in six months period. Patient demographics, procedure, preoperative fasting time, preoperative and postoperative glucose levels were documented. Lactate ringer (LR) solution with % 2 glucose was infused to the patients with preoperative blood glucose level lower than 60 mg/dL, LR solution with % 1 glucose was used for the patients with preoperative blood glucose level between 60-90 mg/dL, LR solution without glucose was used for the patients with preoperative blood glucose level higher than 90 mg/dL.

DETAILED DESCRIPTION:
Lactate ringer (LR) solution with % 2 glucose was infused to the patients with preoperative blood glucose level lower than 60 mg/dL, LR solution with % 1 glucose was used for the patients with preoperative blood glucose level between 60-90 mg/dL, LR solution without glucose was used for the patients with preoperative blood glucose level higher than 90 mg/dL

ELIGIBILITY:
İnclusion criteria;

* 6 months- 12 years old, ASA I-II children
* Undergoing surgery lasting less than four hours were enrolled the study

Exclusion Criteria:

* Diabetes mellitus
* Parenteral nutrition or enteral nutrition
* Patient with metabolic disorders,
* ASA III-IV patients

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
glucose level | perioperative period
  blood glucose level measurement with finger stick monitoring

SECONDARY OUTCOMES:
hyperglysemia or hypoglysemia ratio | perioperative
  blood glucose level measurement with finger stick monitoring